CLINICAL TRIAL: NCT02550639
Title: A Prospective Randomized Study for Predicting Human Cytomegalovirus (hCMV) Infection According to Baseline hCMV-specific T-cell Response in Kidney Transplant Patients (RESPECT)
Brief Title: Prospective, Randomized Study for Predicting Human Cytomegalovirus (hCMV) Infection Based on Baseline hCMV Specific T-cell Response in Kidney Transplant
Acronym: RESPECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ORIOL BESTARD (Other)
Responsible Party: Sponsor-Investigator, ORIOL BESTARD, MD, PhD, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: hCMV2013-RESPECT
Record Dates: First submitted 2015-09-14; First posted 2015-09-15 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: CMV Infection; Kidney Transplantation
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A1-prophylaxis group,positive elispot test (Active Comparator): POSITIVE ELISPOT TEST, PROPHYLAXIS GROUP (CMV PROPHYLAXIS)
  Interventions: Other: BIOMARKER- elispot test
- A2- preemptive group,positive elispot test (Experimental): POSITIVE ELISPOT TEST, PREEMPTIVE GROUP (NO CMV PROPHYLAXIS)
  Interventions: Other: BIOMARKER- elispot test
- B1- prophylaxis group,negative elispot test (Active Comparator): NEGATIVE ELISPOT TEST, PROPHYLAXIS GROUP (CMV PROPHYLAXIS)
  Interventions: Other: BIOMARKER- elispot test
- B2- preemptive group,negative elispot test (Experimental): NEGATIVE ELISPOT TEST, PREEMPTIVE GROUP (NO CMV PROPHYLAXIS)
  Interventions: Other: BIOMARKER- elispot test

INTERVENTIONS:
Other: BIOMARKER- elispot test — ELISPOT TEST

SUMMARY:
The aim of this prospective, randomized study is to assess a subject's immunological status against hCMV before kidney transplantation by an hCMV-specific interferon (INF)-γ ELISPOT technique confirming previous results and establishing their statistical validity in order to determine whether this test could be used routinely in clinical practice to assess the risk of developing hCMV infection after renal transplantation and, ultimately, identify the most effective individual antiviral therapeutic strategy against hCMV.

DETAILED DESCRIPTION:
Human cytomegalovirus (hCMV) is the most common opportunistic pathogen in the first months after solid organ transplantation. Traditionally, hCMV infection in renal transplant patients is indirectly associated with an increased risk of acute rejection, chronic graft dysfunction, graft loss and even increased patient mortality.

The susceptibility of developing hCMV infection is essentially determined by the immune status of the donor and the receptor with regards to the virus, whereby seronegative recipients (IgG) receiving a graft from a seropositive donor (IgG +) are the group of patients with a particularly high risk for developing hCMV infection and disease. In fact, without the administration of a preventative therapy for hCMV, 60 to 70% of this population at risk have an infection (presence of virus in the blood) and up to approximately 20% will develop associated systemic disease (viral invasion of tissues ). Interestingly, the incidence of hCMV infection in patients who are seropositive for the HIV virus and receive a graft is about 20%, increasing to 30% if given cell depletion therapies with polyclonal antibodies administered after transplantation.

There are currently two treatment options to prevent infection by hCMV; One is prophylactic, whereby the antiviral therapy is administered orally for about 90 to 100 days after transplantation in all patients considered at risk (donor IgG+, recipient IgG-) and the second is pre-emptive therapy, in which the presence of virus in the peripheral blood is monitored periodically after transplantation until it appears (at present by polymerase chain reaction (PCR) detection of viral nucleic acids),thus triggering the need for intensive antiviral therapy. When compared with no pharmacological intervention, both therapeutic strategies have demonstrated a significant reduction in the development of hCMV and other herpes virus type diseases, and even a decrease in the incidence of acute graft rejection. However, there are few prospective randomized studies comparing the effectiveness of these two therapeutic alternatives. Recently, a German group prospectively compared the efficacy of prophylactic oral ganciclovir versus intravenous ganciclovir therapy in a group of 148 patients receiving high serological risk renal transplants for hCMV. Interestingly, the group that received prophylactic oral therapy had a higher graft survival at 4 years of follow up (uncensored for death) than the group receiving ganciclovir, suggesting that, despite the administration of intensive intravenous therapy at the time of detection of the virus in the blood, the potential deleterious effect of the virus on the organs during the initial asymptomatic period could explain the benefits of prophylactic therapy from the beginning.

These results have important implications, both clinical and socioeconomic, as they seem to imply the need for systemic prophylaxis to prevent the development of viral infection in all patients currently considered at risk (R -/D +). Moreover, another interesting study which compared primary prophylaxis with oral valganciclovir versus early therapy prevention (pre-emptive therapy) in a large group of kidney transplant recipients with different serologic donor / recipient combinations, showed significantly higher rates of viremia and CMV disease in patients receiving treatment with an incidence of serological CMV infection of up to 53% in serological R + / R + combinations. In this sense, the latest international consensus guidelines indicate that both types of therapy (early and prophylactic) are acceptable, with a degree of moderately high evidence, for groups of seropositive patients receiving a graft from a seropositive donor. The investigator unit has adopted a pre-emptive protocol for the last two years, systematically monitoring viral replication in R + / D + pairs, except in those patients receiving immunosuppressive therapy with Thymoglobulin to whom the investigator assigns a prophylactic treatment with oral valganciclovir for 3 months.This change was introduced 2 years ago before which a prophylactic treatment was given to all R + / R + patients. This change has not led to improved results in terms of prevention of cytomegalic infection.

All such discrepancies among study results examining the efficacy of various therapeutic strategies preventing hCMV could be explained by the poor diagnostic capabilities currently available to identify those patients truly at high risk of developing cytomegalic infection. This is illustrated by the fact that hCMV infection reappears in some patients (15-20%) after transplantation even though they are seropositive (R+) and that, while the majority of patients receiving prophylactic treatment never develop cytomegalic infection after its discontinuation, a small percentage (10-15%) still does, and that, even though 70-80% of seronegative (R-) patients receiving a seropositive graft (R+) will develop post-transplant hCMV infection unless they receive prophylactic treatment, approximately 20-30% never will. All of this leads to important therapeutic contradictions in this field such as that, even though the majority of seropositive recipients will not develop hCMV infection, all of them will still receive an intense and costly monitoring for viremia, and that, although a large majority of patients receiving prophylactic treatment will not develop infection upon treatment discontinuation, continuing such prophylactic antiviral treatment is being proposed across the clinical transplantation community, suggesting that immune surveillance of the risk of developing a post-transplant hCMV infection is currently very poor in clinical practice. It is well established that memory/effector T-cells play a pivotal role in controlling general viral replication and survival, particularly for hCMV. Even though it has been reported that cytotoxic CD8+ T-cells can be activated by a myriad of immunogenic hCMV viral proteins, the predominant and most robust response is directed at the immediate early antigen-1 (IE-1) and phosphoprotein 65 (pp65), which is thought to play a critical role in controlling hCMV replication. Recently published studies suggest that such cellular response is even important for the control and prevention of infection after transplantation.

All such publications, however, refer to the post-transplantation period while patients are under the effects of chronic immunosuppressive therapy and evaluate the T-cell response using assays hardly applicable to routine clinical practice. Even though available, such assays are not used in routine clinical practice to evaluate the hCMV-specific immune response.

One of the most precise functional assays to assess both memory cell and humoral responses under evaluation is the interferon-γ ELISPOT assay. This assay measures antigen-specific memory response frequency by individual cells as they become stimulated.

Recent work in transplantation has established that the detection of highly alloreactive circulating donor-specific T-cells by ELISPOT offers prognostic value when assessing the risk of acute rejection or chronic post-transplant graft dysfunction. Likewise, ELISPOT has been shown to be able to detect highly reactive hCMV-specific T-cells associated with a lower risk of viral infection with both sensitivity and specificity.

The investigator group has recently published that low frequency rates of specific hCMV (IE-1) T-cells before transplantation identify renal transplant recipients at a higher risk of post-transplant hCMV infection with precision, regardless of the therapeutic strategy adopted against hCMV. Remarkably, the same results were observed in patients receiving induction therapy with polyclonal antibodies (Thymoglobuline ®). The investigator thus believes that such an assay approach would allow to identify with precision those patients at risk of developing an infection regardless of their hCMV serology status.

ELIGIBILITY:
Inclusion Criteria:

Adult renal transplant patients fulfilling the following criteria will be included:

1. Subjects must be ≥ 18 years old, with a body weight > 34 kg and of either sex or any race.
2. Subjects must be seropositive for hCMV and must receive a renal graft from a seropositive donor (IgG positive).
3. A pre-transplant blood sample is available from the recipient to carry out an hCMV-specific ELISPOT test.
4. Subjects must be capable of, and willing to provide written informed consent to participate in the study. Subjects unable to provide written informed consent by themselves may be consented through their legal representative.
5. Females of child bearing potential must have a pregnancy test before enrolment and be willing to use a medically acceptable birth control method during the screening period and while they receive study medication.

Exclusion Criteria:

1. An inconclusive hCMV ELISPOT or unavailability of recipient samples.
2. History of type I hypersensitivity reactions or idiosyncratic reactions to ganciclovir (GCV)/valganciclovir (VGCV).
3. Pregnant women.
4. Lactating women.
5. Subjects must not have any clinically significant disease which could interfere with study procedures.
6. Participation in another industry-sponsored clinical study where treatment for CMV is already specified by the study protocol.
7. Patients having received other non-renal transplants.
8. Patients with evidence of active Hepatitis C virus (HCV), Hepatitis B virus (HBV) and/or HIV viral replication.
9. Maintenance immunosuppressive therapy which includes mammalian target of rapamycin (mTOR) inhibitors.
10. Patients requiring desensitization treatment such as plasmapheresis, Campath-1, Rituximab®, Eculizumab® and/or Gammaglobulin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-02; Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
iNCIDENCE OF hCMV INFECTION | 12 MONTHS
  The primary study endpoint is the incidence of hCMV infection in patients receiving Pre-emptive treatment in either group (positive or negative ELISPOT).

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Bestard, MD, PhD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (5):
- Hôpital Erasme- Cliniques Universitaires de Bruxelles,, Brussels, Belgium
- Spain (4):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari de la Vall d'Hebrón, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045
- [Derived] Jarque M, Crespo E, Melilli E, Gutierrez A, Moreso F, Guirado L, Revuelta I, Montero N, Torras J, Riera L, Meneghini M, Taco O, Manonelles A, Paul J, Seron D, Facundo C, Cruzado JM, Gil Vernet S, Grinyo JM, Bestard O. Cellular Immunity to Predict the Risk of Cytomegalovirus Infection in Kidney Transplantation: A Prospective, Interventional, Multicenter Clinical Trial. Clin Infect Dis. 2020 Dec 3;71(9):2375-2385. doi: 10.1093/cid/ciz1209. PMID 32076718